CLINICAL TRIAL: NCT02717117
Title: Reduced Intestinal Motility in Inflammatory Crohn's Disease - Optimisation Studies in Healthy Volunteers
Brief Title: Magnetic Resonance Imaging of Motility in Crohn's 1
Acronym: MIC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H19062014
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Motility; MRI; Gut peptides; Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Feeding (Experimental): Cream of chicken soup (400g) (or mushroom for vegetarians) (Heinz, Wigan, UK) used as a test meal intervention. The nutrient content /100g is: energy (kcal) 51, protein (g) 1.5, carbohydrate (g) 4.7, fat (g) 2.93
  Interventions: Other: Soup meal

INTERVENTIONS:
Other: Soup meal — Soup meal as above

SUMMARY:
Crohn's disease (CD) is becoming more common. One of the main features of this disease is weight loss and malnutrition with symptoms such as tummy aches and bloating. These problems have a strong negative effect on the patients' quality of life but the causes of these problems are not well understood.

Enteroendocrine cells are nutrient sensors in the bowel that secrete special chemicals (called hormones) that control appetite and the movements all the gut. The investigators think that this control mechanism goes wrong in Crohn's patients and they have set off to do more research on this. Looking at the inside work of the gut has always been difficult and at times unpleasant for patients, however recent developments in magnetic resonance imaging (MRI) are allowing the investigators to study the workings of the gut in greater detail and without discomfort for the patients.

Before studying the Crohn's patients it is necessary to run a set of pilot experiments in healthy volunteers using a test meal and subsequent MRI imaging to look at the motion of the gut. This validation stage of the methodology is essential before embarking in more detailed studies in the patients.

DETAILED DESCRIPTION:
Background: Poor nutrition in Crohn's disease (CD) is common but poorly understood. Apart from disease burden and repeated surgery, reduction in appetite might be an aetiological factor.

Enteroendocrine cells (EC) are intraluminal nutrient sensors. They play a pivotal role in orchestrating physiological functions in the gastrointestinal tract. Sensing the nutrient content of the lumen, they secrete multiple peptides and amines that control gut secretory and motor functions. CD patients with small bowel inflammation show increased expression in EC peptides with exaggerated postprandial responses in anorectic EC hormones. This is associated with symptoms of nausea and anorexia, with EC-peptide expression decreasing to normality in remission.

There has been a longstanding interest on the effect of CD on gastric emptying and gastrointestinal motility.

Recent technological advances have allowed us to use magnetic resonance imaging (MRI) to measure both disease activity, intestinal motility and whole gut transit.

Reduced intestinal motility has been recently shown in CD patients with active terminal ileal disease. A significant negative correlation is observed between terminal ileal motility and histological, biochemical and radiological measures of disease activity. Intestinal hypomotility may be observed in proximal unaffected segments of small bowel as well.

An increase in EC activity could potentially lead to altered appetite and symptoms of nausea through delayed gastric emptying and most importantly delayed small bowel transit. This mechanistic link has not been described and present findings have not been correlated to patient symptoms. This work can potentially open a new therapeutic pathway in CD therapy. Optimisation studies in healthy volunteers (HV) are urgently needed.

Aims & Hypothesis: In intestinal inflammation due to CD, the observed up-regulation of fasting and postprandial EC peptides may correlate with a delayed whole gut transit specifically small bowel transit and gastric emptying. This optimization study in HV aims to validate a test meal and optimize themethodology in assessing gastric emptying, small bowel transit and whole gut transit.

Experimental protocol and methods: 15 healthy volunteers will be recruited. Standard MRI exclusion criteria will apply. Volunteers should not have a history of inflammatory bowel disease, history of smoking, a history of bowel resections or any gastric surgery, history of pancreatic insufficiency, thyroid disease, diabetes, protein-pump inhibitor usage or any medication that affects gastric emptying or small bowel transit.

This study will have an open-label design. Subjects will be asked to swallow five MRI marker capsules (20 x 7 mm) at 09:00 am, 24 h before undergoing an MRI scan. The subjects will be asked to fast from 2000 h. They will be asked to fill in a questionnaire to ensure adherence to the study day restrictions.

On the day of the scan, they will only be allowed a small glass of water on waking. They will undergo a baseline fasting scan at 0900 hours (defined at t = -45 min time point), together with a fasting baseline blood sample. At 0925 hours, they will be asked to eat their test meal within a maximum time of 20 min so that at 0945 hours the subjects will undergo a first immediate postprandial scan (defined as t = 0 min). This will be followed with data collection (MRI, questionnaire data and blood samples) time points every 15 min for the first 60 min and every 30 min up to 270 min.

At each time point, the positioning of the subject, setup and data collection will take ~15min. After the first 60 min, at completion of data collection at each time-point, the volunteers will be kept sitting upright in a quiet lounge next to the scanner. At each time point, volunteers will fill a 100mm Visual Analogue Scale (VAS) symptoms questionnaire scoring their feeling of fullness, bloating, distension, abdominal pain/discomfort and nausea. The VAS anchors were from 'not' to 'extremely'. Participants will be given a meal at the end of the study.

MRI scanning will be carried out supine on either a 1.5T or 3.0 T Philips Achieva MRI scanner (Philips Healthcare, Best, The Netherlands) depending on availability. Fasting and post-prandial plasma tests: On the morning of the test, a 10 ml fasting blood sample will be drawn in aprotonin/EDTA tubes (BD-361017, BD Diagnostics, Oxford). Samples will be measured every 45 min to 270 min. Samples will be centrifuged at 4000 rpm for 5 min and stored on ice. Measurement of plasma peptides: All EC peptides (GLP-1, PYY) will be analysed through ELISA techniques (Millipore, UK). Serum CCK will be measured by RIA (Euro Diagnostic Products, Sweden). Total EC plasma peptide response will be presented as per individual time points and compositely as area under the curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body Mass Index (BMI): 18-30 Kg/m2

Exclusion Criteria:

* Patients with a history of inflammatory bowel disease.
* Smokers.
* A history of bowel resections or any gastric surgery.
* History of pancreatic insufficiency, thyroid disease or/and diabetes.
* Protein-pump inhibitor usage or any medication that affects gastric emptying or small bowel transit.
* Any potential participants scoring very highly on the depression scale questionnaire.
* Standard MRI exclusion criteria (e.g. pacemaker).
* Malignant disease
* Stricturing or penetrating disease
* Smoking history
* History of bowel resections or any gastric surgery
* Significant cardiovascular or respiratory disease
* Current Infection
* Neurological or cognitive impairment
* Significant physical disability
* Significant hepatic disease or renal failure
* Subjects currently (or in the last three months) participating in another research project
* pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Small bowel motility | From fasting baseline to 270 min postprandially
  MRI small bowel motility index (arbitrary units)

SECONDARY OUTCOMES:
Gall bladder contraction | From fasting baseline to 60 min postprandially
  Gall bladder contraction from MRI images
Gastric volumes | From fasting baseline to 150 min postprandially
  Gastric emptying from gastric volumes time courses
Small bowel water content | From fasting baseline to 270 min postprandially
  Small bowel water content from MRI images
Whole gut transit | 24 hours after ingestion of the MRI transit capsules
  Whole gut transit weighted average position scores
Plasma GLP-1 | From fasting baseline to 270 min postprandially
  Postprandial GLP-1 peptide response
Plasma PYY | From fasting baseline to 270 min postprandially
  Postprandial PYY peptide response
Plasma CCK | From fasting baseline to 270 min postprandially
  Postprandial CCKpeptide response
Satiety | From fasting baseline to 270 min postprandially
  Satiety VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Moran, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre, QMC Campus, Nottingham University Hospitals, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No